CLINICAL TRIAL: NCT00304694
Title: Whole-Body 18F-FDG PET in Evaluating Induction Chemotherapeutic Response for Locally Advanced Nasopharyngeal Cancer Patients and Correlating With Histopathology: a Prospective Study
Brief Title: Whole-Body 18F-FDG PET in Induction Chemotherapeutic Response for Advanced NPC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 940601
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2006-03-20 (Estimated); Status verified 2006-03

CONDITIONS: Nasopharyngeal Cancer
Keywords: NPC; Induction chemotherapy; Therapeutic response; 18F-FDG PET
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
18F-FDG PET, a whole-body imaging technology based on glucose metabolism, can effectively detect subclinical and clinical therapeutic responses at stages that are earlier than those detected by conventional approaches.

We propose to conduct a prospective study to evaluate therapeutic response using 18F-FDG PET before and after induction chemotherapy for locally advanced NPC patients.

DETAILED DESCRIPTION:
In order to improve locoregional control and to eradicate micrometastases for patients with locally advanced nasopharyngeal carcinoma (NPC), induction chemotherapy followed by concurrent chemoradiotherapy has been the preferred therapeutic approach.Although it would be of great advantage to identify non-responder during or immediately after therapy to formulate an alternative treatment strategy, non-invasive methods for early evaluation of therapeutic response for advanced NPC patients have not been fully evaluated. Decrease of tumor volume in anatomical images and relief of symptoms in clinical follow-up have been used in many conventional approaches to evaluate the effectiveness of therapy. However, an effective therapy could very well have resulted in early subclinical alterations in tumor physiology and biochemistry. These alterations may have occurred long before changes in the tumor mass become apparent. Thus therapeutic effect may not be assessed accurately using the conventional anatomical imaging studies, such as CT and MRI.Recent studies have shown that 18F-FDG PET, a whole-body imaging technology based on glucose metabolism, can effectively detect subclinical and clinical therapeutic responses at stages that are earlier than those detected by conventional approaches.We therefore propose to conduct a prospective study to evaluate therapeutic response using 18F-FDG PET before and after induction chemotherapy for locally advanced NPC patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed locally advanced NPC patients who are receiving induction chemotherapy for treatment

Exclusion Criteria:

* age below 18 year old
* pregnancy women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Ruoh-Fang Yen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan